CLINICAL TRIAL: NCT02409368
Title: An Open-Label, Multicenter Clinical Trial With Nivolumab (BMS-936558) Monotherapy in Subjects With Advanced or Metastatic Squamous Cell (Sq) Non-Small Cell Lung Cancer (NSCLC) Who Have Received at Least One Prior Systemic Regimen for the Treatment of Stage IIIb/IV SqNSCLC
Acronym: Checkmate 171
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CA209-171; 2014-001285-10 (EudraCT Number)
Record Dates: First submitted 2015-04-01; First posted 2015-04-06 (Estimated); Results first posted 2021-07-29 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cohort A: Treatment - Nivolumab (Experimental): Nivolumab IV infusion
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab

SUMMARY:
The purpose of the study is to determine the occurrence of high-grade (CTCAE v4.0 Grades 3-4), treatment-related, select adverse events in patients with advanced or metastatic Squamous Cell Non-Small Cell Lung Cancer (SqNSCLC) with progression of disease during or after at least 1 systemic therapy.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* ECOG Status: PS 0-1 & PS 2
* Subjects with histologically or cytologically-documented SqNSCLC
* Subjects must have experienced disease progression or recurrence during or after one prior platinum doublet-based chemotherapy regimen
* Subjects must have evaluable disease by CT or MRI per RECIST 1.1 criteria
* Subjects with treated or asymptomatic CNS metastases
* Prior palliative radiotherapy must have been completed at least 14 days prior to study drug administration
* Prior lines of antineoplastic therapy, including hemotherapy, hormonal therapy, immunotherapy, surgical resection of lesions, non-palliative radiation therapy, or standard or investigational agents for treatment of NSCLC, must be completed 28 days prior to the first dose of nivolumab
* Males and Females, ages 18 or older

Exclusion Criteria:

* Subjects with untreated, symptomatic CNS metastases
* Subjects with carcinomatous meningitis
* Subjects with active, known or suspected autoimmune disease.
* Subjects who received prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways) or who have previously taken part in a randomized BMS clinical trial for nivolumab or ipilimumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 812 (Actual)
Dates: Start 2015-04-29 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2021-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (90):
- Austria (3):
  - Local Institution - 0002, Wels, Upper Austria
  - Local Institution - 0003, Salzburg
  - Local Institution - 0005, Vienna
- Denmark (3):
  - Local Institution - 0173, Odense, Region Syddanmark
  - Local Institution - 0021, Aalborg
  - Local Institution - 0020, Herlev
- Finland (2):
  - Local Institution - 0022, Oulu, North Ostrobothnia
  - Local Institution - 0023, Pori
- Greece (5):
  - Local Institution - 0051, Athens
  - Local Institution - 0052, Heraklion
  - Local Institution - 0177, Nea Kifisia Athens
  - Local Institution - 0148, Pátrai
  - Local Institution - 0147, Thessaloniki
- Hungary (4):
  - Local Institution - 0054, Pécs, Baranya
  - Local Institution - 0053, Budapest
  - Local Institution - 0347, Budapest
  - Local Institution - 0178, Debrecen
- Ireland (3):
  - Local Institution - 0056, Dublin
  - Local Institution - 0058, Galway
  - Local Institution - 0349, Tullamore, Offaly
- Poland (6):
  - Local Institution - 0087, Poznan, Greater Poland Voivodeship
  - Local Institution - 0158, Gliwice, Silesian Voivodeship
  - Local Institution - 0184, Zabrze, Silesian Voivodeship
  - Local Institution - 0086, Gdansk
  - Local Institution - 0088, Lodz
  - Local Institution - 0089, Warsaw
- Portugal (6):
  - Local Institution - 0094, Coimbra
  - Local Institution - 0093, Lisbon
  - Local Institution - 0090, Lisbon
  - Local Institution - 0092, Porto
  - Local Institution - 0091, Porto
  - Local Institution - 0159, Porto
- Romania (6):
  - Local Institution - 0192, Oradea, Bihor County
  - Local Institution - 0098, Cluj-Napoca, Cluj
  - Local Institution - 0187, Timișoara, Timiș County
  - Local Institution - 0095, Bucharest
  - Local Institution - 0096, Bucharest
  - Local Institution - 0097, Cluj-Napoca
- Russia (3):
  - Local Institution - 0100, Saint Petersburg, Leningradskaya Oblast'
  - Local Institution - 0160, Moscow, Moscow
  - Local Institution - 0099, Saint Petersburg, Sankt-Peterburg
- Spain (21):
  - Local Institution - 0109, Santander, Cantabria
  - Local Institution - 0337, Oviedo, Principality of Asturias
  - Local Institution - 0107, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Local Institution - 0104, A Coruña
  - Local Institution - 0119, Alicante
  - Local Institution - 0162, Barcelona
  - Local Institution - 0112, Barcelona
  - Local Institution - 0111, Barcelona
  - Local Institution - 0110, Barcelona
  - Local Institution - 0108, Burgos
  - Local Institution - 0103, Granada
  - Local Institution - 0114, Madrid
  - Local Institution - 0117, Madrid
  - Local Institution - 0116, Madrid
  - Local Institution - 0105, Madrid
  - Local Institution - 0106, Málaga
  - Local Institution - 0113, Palma de Mallorca
  - Local Institution - 0118, Seville
  - Local Institution - 0161, Valencia
  - Local Institution - 0102, Valencia
  - Local Institution - 0163, Zaragoza
- Sweden (6):
  - Local Institution - 0346, Stockholm, Stockholm County
  - Local Institution - 0193, Gothenburg, Västra Götaland County
  - Local Institution - 0348, Linköping
  - Local Institution - 0342, Lund
  - Local Institution - 0120, Stockholm
  - Local Institution - 0339, Örebro, Örebro County
- United Kingdom (22):
  - Local Institution - 0345, Aberdeen, Aberdeen CITY
  - Local Institution - 0127, London, Greater London
  - Local Institution - 0191, Manchester, Greater Manchester
  - Local Institution - 0131, Southampton, Hampshire
  - Local Institution - 0128, Maidstone, Kent
  - Local Institution - 0195, Glasgow, Lanarkshire
  - Local Institution - 0132, Preston, Lancashire
  - Local Institution - 0167, Leicester, Leicestershire
  - Local Institution - 0196, Sutton, Surrey
  - Local Institution - 0171, Bebington
  - Local Institution - 0340, Bodelwyddan, Rhyl
  - Local Institution - 0344, Bradford
  - Local Institution - 0190, Bristol
  - Local Institution - 0133, Cardiff
  - Local Institution - 0126, Cottingham
  - Local Institution - 0165, London
  - Local Institution - 0169, London
  - Local Institution - 0194, Northwood
  - Local Institution - 0166, Plymouth
  - Local Institution - 0124, Sheffield
  - Local Institution - 0189, Sutton
  - Local Institution - 0338, West Midlands

REFERENCES:
- [Derived] Felip E, Ardizzoni A, Ciuleanu T, Cobo M, Laktionov K, Szilasi M, Califano R, Carcereny E, Griffiths R, Paz-Ares L, Duchnowska R, Garcia MA, Isla D, Jassem J, Appel W, Milanowski J, Van Meerbeeck JP, Wolf J, Li A, Acevedo A, Popat S. CheckMate 171: A phase 2 trial of nivolumab in patients with previously treated advanced squamous non-small cell lung cancer, including ECOG PS 2 and elderly populations. Eur J Cancer. 2020 Mar;127:160-172. doi: 10.1016/j.ejca.2019.11.019. Epub 2020 Feb 3. PMID 32028209
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant was ECOG PS 3 and thus outside the scope of the protocol and excluded from analysis.
  There were 2 ECOG classification periods during the course of this study. The population from the first was used in the Primary Outcome Measure analysis. The population from the second was used in the Baseline Characteristics, Secondary Outcome Measures, and Adverse Event analysis. 1 participant was lost from the Primary Completion ECOG Classification that was accounted for at Study Completion.
Groups:
- ECOG (PS0): ECOG Performance Status 0
  Nivolumab 3 mg/kg as a 60- minute IV infusion every 2 weeks
- ECOG (PS1): ECOG Performance Status 1
  nivolumab 3 mg/kg as a 60- minute IV infusion every 2 weeks
- ECOG Performance Status 2: Nivolumab 3 mg/kg as a 60-minute IV infusion every 2 weeks
- ECOG (PS3): ECOG Performance Status 3
  nivolumab 3 mg/kg as a 60- minute IV infusion every 2 weeks
Period: Original Classification
Arm/Group | ECOG (PS0) | ECOG (PS1) | ECOG Performance Status 2 | ECOG (PS3)
Started | 173 | 534 | 103 | 1
Completed | 173 | 534 | 103 | 1
Not Completed | 0 | 0 | 0 | 0
Period: ECOG Reclassification
Arm/Group | ECOG (PS0) | ECOG (PS1) | ECOG Performance Status 2 | ECOG (PS3)
Started | 172 | 537 | 102 | 1
Completed | 0 | 0 | 0 | 0
Not Completed | 172 | 537 | 102 | 1
Not completed — Adverse event unrelated to study drug | 17 | 49 | 12 | 0
Not completed — Death | 1 | 5 | 0 | 0
Not completed — Disease Progression | 113 | 382 | 70 | 1
Not completed — Lost to Follow-up | 1 | 5 | 0 | 0
Not completed — Maximum clinical benefit | 6 | 5 | 0 | 0
Not completed — Poor/non-compliance | 0 | 3 | 2 | 0
Not completed — Study drug toxicity | 17 | 42 | 7 | 0
Not completed — Participant no longer meets study criteria | 3 | 8 | 3 | 0
Not completed — Participant request to discontinue study treatment | 6 | 6 | 2 | 0
Not completed — Participant withdrew consent | 2 | 3 | 4 | 0
Not completed — Other Reasons | 5 | 26 | 2 | 0
Not completed — Administrative reason by sponsor | 1 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are listed for all treated participants from the Study Completion ECOG Classification.
Groups:
- Total: Total of all reporting groups
Arm/Group | ECOG (PS0) | ECOG (PS1) | ECOG Performance Status 2 | ECOG (PS3) | Total
Number analyzed (Participants) | 172 | 537 | 102 | 1 | 812
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.6 (8.28) | 66.1 (8.27) | 67.9 (7.29) | 71 (NA) — Standard deviation not calculated due to insufficient data | 65.8 (8.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 111 | 22 | 1 | 171
  Male | 135 | 426 | 80 | 0 | 641
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 37 | 11 | 0 | 61
  Not Hispanic or Latino | 159 | 500 | 91 | 1 | 751
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 0 | 0 | 3
  White | 165 | 530 | 102 | 1 | 798
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 2 | 0 | 0 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With High Grade (Grade 3, 4 and 5) Treatment Related Select Adverse Events
Description: The total number of participants with high grade treatment related select adverse events.
Time Frame: From first dose to time of analysis of primary endpoint (approximately up to 34 months)
Population: All Treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | ECOG (PS0) | ECOG (PS1) | ECOG Performance Status 2
Number analyzed (Participants) | 173 | 534 | 103
Participants
  Skin | 1 | 7 | 0
  Gastrointestinal | 1 | 10 | 0
  Endocrine | 4 | 3 | 0
  Hepatic | 3 | 11 | 2
  Pulmonary | 2 | 5 | 0
  Renal | 0 | 3 | 1
  Hypersensitivity/ Infusion reaction | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With High Grade Select Adverse Events
Description: The total number of participants with high grade select adverse events. High grade is defined as Common Terminology Criteria for Adverse Events (CTCAE) v4.0 Grades 3-4. An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation subject administered study drug and that does not necessarily have a causal relationship with this treatment. Select AEs include Pulmonary toxicity, Gastrointestinal toxicity (diarrhea or colitis, Endocrinopathies, Hepatotoxicity (including asymptomatic LFT elevations), Renal toxicity, Skin toxicity, and Neurological toxicity.
Time Frame: From first dose up to 100 days post last dose (up to 76 months)
Population: All treated participants with ECOG PS Grade 0-2
Measure: Count of Participants; unit: Participants
Arm/Group | ECOG (PS0) | ECOG (PS1) | ECOG Performance Status 2
Number analyzed (Participants) | 172 | 537 | 102
Participants
  Skin | 2 | 7 | 0
  Gastrointestinal | 1 | 11 | 0
  Endocrine | 5 | 4 | 0
  Hepatic | 6 | 19 | 3
  Pulmonary | 3 | 9 | 1
  Renal | 0 | 7 | 1
  Hypersensitivity/ Infusion reaction | 0 | 0 | 1

3. Secondary Outcome: Median Time to Onset of Any Grade Select Adverse Events
Description: Median Time to onset of any grade select adverse events reported up to 100 days after last dose. An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation subject administered study drug and that does not necessarily have a causal relationship with this treatment. Select AEs include Pulmonary toxicity, Gastrointestinal toxicity (diarrhea or colitis, Endocrinopathies, Hepatotoxicity (including asymptomatic LFT elevations), Renal toxicity, Skin toxicity, and Neurological toxicity.
Time Frame: From first dose up to 100 days post last dose (up to approximately 65 months)
Population: All treated participants with ECOG PS Grade 0-2
Measure: Median (Full Range); unit: Weeks
Arm/Group | ECOG (PS0) | ECOG (PS1) | ECOG Performance Status 2
Number analyzed (Participants) | 172 | 537 | 102
Weeks
  Endrocrine: number analyzed (Participants) | 42 | 62 | 7
  Endrocrine | 12.79 [4.0 to 121.6] | 10.14 [1.9 to 165.1] | 19.86 [6.1 to 55.4]
  Gastrointestinal: number analyzed (Participants) | 25 | 101 | 17
  Gastrointestinal | 11.71 [0.1 to 88.0] | 8.86 [0.1 to 228.1] | 6.00 [0.3 to 64.3]
  Hepatic: number analyzed (Participants) | 20 | 58 | 11
  Hepatic | 26.64 [1.4 to 234.1] | 11.43 [2.0 to 90.1] | 8.14 [2.0 to 88.1]
  Pulmonary: number analyzed (Participants) | 13 | 34 | 4
  Pulmonary | 33.43 [7.4 to 169.4] | 11.50 [0.6 to 166.0] | 3.93 [0.1 to 26.3]
  Renal: number analyzed (Participants) | 13 | 51 | 7
  Renal | 28.86 [4.1 to 129.9] | 22.71 [0.1 to 246.0] | 10.29 [1.4 to 52.9]
  Skin: number analyzed (Participants) | 31 | 132 | 19
  Skin | 12.14 [0.1 to 92.1] | 7.86 [0.1 to 200.1] | 14.71 [2.1 to 81.7]
  Hypersensitivity/Infusion Reaction: number analyzed (Participants) | 2 | 12 | 4
  Hypersensitivity/Infusion Reaction | 1.93 [1.7 to 2.1] | 2.21 [0.3 to 20.3] | 2.14 [2.1 to 28.6]

4. Secondary Outcome: Median Time to Resolution of Any Grade Select Adverse Events
Description: Median time to resolution of any grade select adverse events reported up to 100 days after last dose. An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation subject administered study drug and that does not necessarily have a causal relationship with this treatment. Select AEs include Pulmonary toxicity, Gastrointestinal toxicity (diarrhea or colitis, Endocrinopathies, Hepatotoxicity (including asymptomatic LFT elevations), Renal toxicity, Skin toxicity, and Neurological toxicity.
Time Frame: From first dose to up to 100 days post last dose (up to approximately 45 months)
Population: All treated participants with ECOG PS Grade 0-2
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | ECOG (PS0) | ECOG (PS1) | ECOG Performance Status 2
Number analyzed (Participants) | 172 | 537 | 102
Weeks
  Endrocrine: number analyzed (Participants) | 42 | 62 | 7
  Endrocrine | NA [109.00 to NA] — Median and upper limit not reached due to insufficient number of events | 169.43 [17.86 to NA] — Upper limit not reached due to insufficient number of events | NA [6.14 to NA] — Median and upper limit not reached due to insufficient number of events
  Gastrointestinal: number analyzed (Participants) | 25 | 101 | 17
  Gastrointestinal | 2.86 [0.43 to 5.14] | 2.00 [1.00 to 3.00] | 2.00 [0.43 to 5.71]
  Hepatic: number analyzed (Participants) | 20 | 57 | 11
  Hepatic | 4.57 [2.57 to 6.14] | 7.71 [4.86 to 17.14] | 3.57 [2.14 to 8.14]
  Pulmonary: number analyzed (Participants) | 13 | 34 | 4
  Pulmonary | 3.00 [1.43 to NA] — Upper limit not reached due to insufficient number of events | 4.29 [2.14 to 6.00] | 2.29 [1.00 to NA] — Upper limit not reached due to insufficient number of events
  Renal: number analyzed (Participants) | 13 | 51 | 7
  Renal | 10.14 [2.14 to NA] — Upper limit not reached due to insufficient number of events | 6.14 [2.29 to 25.14] | 59.14 [0.57 to 59.14]
  Skin: number analyzed (Participants) | 31 | 132 | 19
  Skin | NA [13.57 to NA] — Median and upper limit not reached due to insufficient number of events | 15.43 [8.71 to 52.86] | 5.71 [2.00 to NA] — Upper limit not reached due to insufficient number of events
  Hypersensitivity/Infusion Reaction: number analyzed (Participants) | 2 | 12 | 4
  Hypersensitivity/Infusion Reaction | 1.14 [0.14 to 2.14] | 0.14 [0.14 to 4.43] | 0.14 [0.14 to 0.71]

5. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) is defined as the time from first dosing date to the date of death. A subject who has not died will be censored at last known date alive. OS will be followed continuously while subjects are on treatment and every 3 months via in-person or phone contact after subjects discontinue the study drug.
Time Frame: From the first dosing up to the date of death (up to approximately 76 months)
Population: All treated participants with ECOG PS Grade 0-2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | ECOG (PS0) | ECOG (PS1) | ECOG Performance Status 2
Number analyzed (Participants) | 172 | 537 | 102
Months | 12.1 [9.9 to 13.4] | 10.3 [9.3 to 11.3] | 5.2 [3.0 to 7.6]

6. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of subjects with a best overall response (BOR) of confirmed complete response (CR) or partial response (PR). CR is defined as the disappearance of all target lesions; PR is defined by at least a 30% decrease in the sum of the longest diameter of target lesions. ORR as assessed by the investigator will be reported.
Time Frame: From first dose up to last dose (up to approximately 76 months)
Population: All response evaluable participants
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | ECOG (PS0) | ECOG (PS1) | ECOG Performance Status 2
Number analyzed (Participants) | 150 | 456 | 64
Percentage | 8.0 [4.2 to 13.6] | 11.0 [8.2 to 14.2] | 1.6 [0.0 to 8.4]

7. Post Hoc Outcome: Number of Participants With High Grade (Grade 3, 4 and 5) Treatment Related Select Adverse Events - Extended Collection
Description: The total number of participants with high grade treatment related select adverse events. High grade is defined as Common Terminology Criteria for Adverse Events (CTCAE) v4.0 Grades 3-4 or 5. An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation subject administered study drug and that does not necessarily have a causal relationship with this treatment. Select AEs include Pulmonary toxicity, Gastrointestinal toxicity (diarrhea or colitis, Endocrinopathies, Hepatotoxicity (including asymptomatic LFT elevations), Renal toxicity, Skin toxicity, and Neurological toxicity.
  Note: This outcome measure represents an updated version of the primary endpoint to include additional data collection that has occurred after the primary completion date.
Time Frame: From first dose to up to 100 days post last dose (up to approximately 76 months)
Population: All treated participants with ECOG PS Grade 0-2
Measure: Count of Participants; unit: Participants
Arm/Group | ECOG (PS0) | ECOG (PS1) | ECOG Performance Status 2
Number analyzed (Participants) | 172 | 537 | 102
Participants
  Skin | 2 | 7 | 0
  Gastrointestinal | 1 | 10 | 0
  Hepatic | 4 | 12 | 2
  Pulmonary | 2 | 6 | 0
  Renal | 0 | 3 | 1
  Hypersensitivity/ Infusion reaction | 0 | 0 | 0
  Endocrine | 4 | 3 | 0

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their enrollment to study completion, (up to approximately 73 months). SAEs and Other AEs were assessed from first dose to 100 days following last dose (up to approximately 76 months)
Groups:
- ECOG Performance Status 0; ECOG Performance Status 1; ECOG Performance Status 2; ECOG Performance Status 3: Nivolumab 3 mg/kg as a 60-minute IV infusion every 2 weeks
Arm/Group | ECOG Performance Status 0 | ECOG Performance Status 1 | ECOG Performance Status 2 | ECOG Performance Status 3
All-Cause Mortality (participants affected / at risk) | 131/172 | 446/537 | 90/102 | 1/1
Serious Adverse Events (participants affected / at risk) | 115/172 | 375/537 | 84/102 | 1/1
Other Adverse Events (participants affected / at risk) | 149/172 | 472/537 | 86/102 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ECOG Performance Status 0 (N=172) | ECOG Performance Status 1 (N=537) | ECOG Performance Status 2 (N=102) | ECOG Performance Status 3 (N=1)
Anaemia (Blood and lymphatic system disorders) | 2 | 6 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 2 | 2 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 3 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 3 | 1 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0 | 0 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 1 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0
Mitral valve prolapse (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 3 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 3 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 3 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 2 | 1 | 0 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Hypophysitis (Endocrine disorders) | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 2 | 2 | 0 | 0
Thyroiditis (Endocrine disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Autoimmune colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Colitis microscopic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 7 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 4 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oesophageal rupture (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 3 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Asthenia (General disorders) | 0 | 2 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Death (General disorders) | 0 | 1 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 1
General physical health deterioration (General disorders) | 1 | 4 | 1 | 0
Hernia obstructive (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 4 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 8 | 0 | 0
Sudden cardiac death (General disorders) | 0 | 1 | 1 | 0
Sudden death (General disorders) | 1 | 4 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1 | 2 | 0
Biliary tract disorder (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Bacterial diarrhoea (Infections and infestations) | 0 | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0
Biliary sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 4 | 9 | 1 | 0
Bronchitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 2 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium colitis (Infections and infestations) | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 2 | 0
H1N1 influenza (Infections and infestations) | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 2 | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 3 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 5 | 21 | 5 | 0
Mediastinitis (Infections and infestations) | 0 | 0 | 1 | 0
Meningitis aseptic (Infections and infestations) | 0 | 1 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 20 | 41 | 10 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia fungal (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 1 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 3 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 11 | 25 | 3 | 0
Sepsis (Infections and infestations) | 3 | 7 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 5 | 1 | 0
Vulval abscess (Infections and infestations) | 0 | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0
Liver function test increased (Investigations) | 0 | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 12 | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 3 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 59 | 206 | 58 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5 | 2 | 0
Brain oedema (Nervous system disorders) | 0 | 2 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 2 | 1 | 0
Coma (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 2 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 2 | 0 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Monoparesis (Nervous system disorders) | 0 | 1 | 0 | 0
Motor dysfunction (Nervous system disorders) | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 3 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 2 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 3 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 2 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 2 | 0 | 0
Mania (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 4 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 2 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 4 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 5 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 28 | 10 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7 | 11 | 3 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 10 | 2 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 15 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 10 | 1 | 0
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1 | 0
Embolism (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0 | 0
Superior vena cava occlusion (Vascular disorders) | 1 | 2 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 4 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ECOG Performance Status 0 (N=172) | ECOG Performance Status 1 (N=537) | ECOG Performance Status 2 (N=102) | ECOG Performance Status 3 (N=1)
Anaemia (Blood and lymphatic system disorders) | 23 | 97 | 21 | 1
Hypothyroidism (Endocrine disorders) | 25 | 37 | 6 | 0
Constipation (Gastrointestinal disorders) | 18 | 80 | 16 | 0
Diarrhoea (Gastrointestinal disorders) | 26 | 100 | 16 | 0
Nausea (Gastrointestinal disorders) | 20 | 71 | 16 | 0
Vomiting (Gastrointestinal disorders) | 9 | 34 | 9 | 1
Asthenia (General disorders) | 30 | 131 | 15 | 0
Fatigue (General disorders) | 40 | 121 | 25 | 1
Non-cardiac chest pain (General disorders) | 6 | 34 | 5 | 0
Oedema peripheral (General disorders) | 7 | 30 | 14 | 1
Pyrexia (General disorders) | 9 | 49 | 8 | 0
Lower respiratory tract infection (Infections and infestations) | 18 | 51 | 7 | 0
Respiratory tract infection (Infections and infestations) | 10 | 37 | 6 | 0
Upper respiratory tract infection (Infections and infestations) | 10 | 29 | 2 | 0
Alanine aminotransferase increased (Investigations) | 12 | 30 | 5 | 0
Aspartate aminotransferase increased (Investigations) | 15 | 28 | 5 | 0
Blood creatinine increased (Investigations) | 9 | 34 | 5 | 0
Weight decreased (Investigations) | 8 | 42 | 7 | 0
Decreased appetite (Metabolism and nutrition disorders) | 24 | 147 | 24 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 6 | 39 | 6 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 11 | 27 | 5 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 52 | 7 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 46 | 7 | 1
Headache (Nervous system disorders) | 10 | 36 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 44 | 134 | 19 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 44 | 167 | 28 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 11 | 47 | 10 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 58 | 10 | 0
Rash (Skin and subcutaneous tissue disorders) | 10 | 39 | 5 | 0
Hyperthyroidism (Endocrine disorders) | 13 | 18 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 28 | 3 | 0
Stomatitis (Gastrointestinal disorders) | 5 | 14 | 7 | 0
Chest pain (General disorders) | 10 | 24 | 1 | 0
Influenza like illness (General disorders) | 3 | 4 | 2 | 1
Peripheral swelling (General disorders) | 2 | 8 | 2 | 1
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 11 | 15 | 1 | 0
Oral candidiasis (Infections and infestations) | 4 | 26 | 3 | 1
Oral fungal infection (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 11 | 24 | 5 | 0
Tooth infection (Infections and infestations) | 2 | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 7 | 20 | 6 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 | 24 | 7 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 25 | 6 | 1
Dizziness (Nervous system disorders) | 3 | 28 | 8 | 0
Seizure (Nervous system disorders) | 0 | 2 | 0 | 1
Anxiety (Psychiatric disorders) | 9 | 12 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10 | 22 | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 26 | 6 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 26 | 6 | 0
Hypertension (Vascular disorders) | 12 | 19 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2018-09-10): https://cdn.clinicaltrials.gov/large-docs/68/NCT02409368/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/68/NCT02409368/SAP_001.pdf